CLINICAL TRIAL: NCT04557722
Title: The Newly Reported (0-90°) Versus (0-30°) Biplanar Fluoroscopic Puncture Technique for Percutaneous Nephrolithotomy: Prospective Randomized Study
Brief Title: The Newly Reported (0-90°) Versus (0-30°) Biplanar Fluoroscopic Puncture Technique in PCNL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed Zakaria Ali Ibrahim Alshahawy, Principal Investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: New 0-90° Vs 0-30° in PCNL
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Nephrolithotomy, Percutaneous; Kidney Stone; PCNL
Keywords: PCNL; 0-30º Biplanar; new 0-90º; PCNL puncture techniques; 090 PCNL; 030 PCNL
MeSH Terms: conditions — Kidney Calculi | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: 0-30° technique. (Active Comparator): Procedure: 0-30° Biplanar Fluoroscopic Puncture Technique for Percutaneous Nephrolithotomy.
  Interventions: Procedure: 0-30° Biplanar Fluoroscopic Puncture Techniques for Percutaneous Nephrolithotomy
- Group 2: new 0-90° technique. (Active Comparator): Procedure: new 0-90° Fluoroscopic Puncture Technique for Percutaneous Nephrolithotomy.
  Interventions: Procedure: New 0-90° Fluoroscopic Puncture Techniques for Percutaneous Nephrolithotomy

INTERVENTIONS:
Procedure: 0-30° Biplanar Fluoroscopic Puncture Techniques for Percutaneous Nephrolithotomy — after retrograde instillation of contrast through the ureteric catheter; the puncture of the desired calyx by using the 0-30 degree technique of C-Arm.
  Arms: Group 1: 0-30° technique.
Procedure: New 0-90° Fluoroscopic Puncture Techniques for Percutaneous Nephrolithotomy — after retrograde instillation of contrast through the ureteric catheter; the puncture of the desired calyx by using the 0-90 degree technique of C-Arm.
  Arms: Group 2: new 0-90° technique.

SUMMARY:
To analyze and compare the puncture success rate, puncture fluoroscopy time and intraoperative puncture complications of two different puncture techniques; fluoroscopic bi-planar (0-30º) versus newly reported bi-planar (0-90º) technique in PCNL.

DETAILED DESCRIPTION:
Nephrolithiasis is one of the most common urological diseases, it is a widespread and challenging issue for both patients and healthcare systems. It is responsible for a significant financial and psychological burden, with an increased incidence of disease. The EAU (European Association of Urology) Guidelines recommend percutaneous nephrolithotomy in patients with kidney stones >2 cm.

The most crucial step of the procedure is the precise puncture of the caliceal system. This can be accomplished by the use of fluoroscopy, ultrasound, or the combination of both and new other imaging modalities techniques. Among them, Fluoroscopy is the most common method for conducting the percutaneous puncture by urologists worldwide using multiple mono-planar or bi-planar fluoroscopic techniques.

However, all fluoroscopic approaches face the same limitation, which is the difficult interpretation of the three-dimensional renal anatomy based on the two-dimensional X-ray information. Another disadvantage is the amount of fluoroscopic radiation used. Surgeons, assistants, nurses and patients, however, all have to accept various levels of radiation exposure. Numerous researches have revealed that it is still harmful to the human body who is exposed to radiation frequently, although under the aegis of protective aprons and thyroid shields, thus the application is affected to varying degrees.

Fluoroscopic bi-planar techniques provide better information about the depth and direction of the collecting system than mono-planar methods. The most popular bi-planar methods described in the literature are the triangulation (0-30º), the "bull´s eye" technique and the less known bi-planar technique (The 0-90º technique) described by Dr. Paul Escovar. A newly published (0-90º) technique by Braulio O Manzo et al to increase the accuracy of calculating the needle path to the exact calyx depth and decreases its radiation exposure.

In the current study, the investigator aimed to compare two different renal access techniques; fluoroscopic 0-30 and modified 0-90 technique regarding success rate, fluoroscopy time and intraoperative puncture complications.

ELIGIBILITY:
Inclusion Criteria:

* A patient over 18 years old.
* Renal stone 2 cm or greater.

Exclusion Criteria:

* A patient < 18 years old.
* Congenital anomalies of the kidney: horseshoe kidney, malrotated kidney, pelvic ectopic kidney.
* Patient with obvious spinal deformity.
* Coagulopathies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The puncture success rate and number of attempts | intraoperative
  percentage of patients in whom the renal puncture achieving desired calyx (evaluated by adequate introduction of the guidewire, bright urine output and stone accessibility).

SECONDARY OUTCOMES:
The Puncture fluoroscopy screening time | intraoperative
  assessed on the monitor of C-Arm.
Intraoperative puncture complications | intraoperative
  1. Dye Extravasation:
     * Mild extravasation of contrast.
     * Significant extravasation which obscure important anatomical detail and making accurate needle redirection impossible.
  2. Puncture failure rate: when puncture failed on achieving desired calyx, conversion into another puncture technique will be made.
  3. Bleeding:
     * Mild intraoperative bleeding.
     * Significant bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elshazly, MD, Study Director — Menoufia University; Mohamed Kamal Omar, MD, Study Director — Menoufia University; Eid El Sherif, MD, Study Director — Menoufia University; Mohamed Aziz, MD, Study Director — Menoufia University
Locations (1):
- MenoufiaU, Menoufia, Shebin El-kom, Egypt

IPD SHARING:
Plan to Share IPD: No